CLINICAL TRIAL: NCT00289341
Title: A Phase I/II Study of Autologous Dendritic Cells Pulsed With Apoptotic Tumor Cells (DC/LNCaP) Administered Subcutaneously to Prostate Cancer Patients.
Brief Title: Safety and Effectiveness of a Vaccine for Prostate Cancer That Uses Each Patients' Own Immune Cells.
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Rockefeller University (Other)
Responsible Party: Principal Investigator, Robert Darnell, Principal Investigator, Rockefeller University
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: RDA 0466
Record Dates: First submitted 2006-02-07; First posted 2006-02-09 (Estimated); Results first posted 2013-01-08 (Estimated); Last update posted 2013-01-18 (Estimated); Status verified 2013-01

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Placebo (Placebo Comparator): 12 patients in the placebo Arm for 8 weeks followed by DC/LNCAP, DC/LNCaP-M1 and DC/KLH immunizations over 8 weeks.
  Interventions: Biological: vaccine vehicle only
- DC/LNCaP (Experimental): 12 patients, receiving DC/LNCaP, DC/LNCaP-M1 and DC/KLH immunizations over 8 weeks
  Interventions: Biological: DC/LNCaP

INTERVENTIONS:
Biological: vaccine vehicle only — Subcutaneous injection of vaccine vehicle only (5% DMSO in normal saline), followed by cross-over to Arm 1 design.
  Arms: Placebo
Biological: DC/LNCaP — Subcutaneous injection of DC/LNCaP, DC/LNCaP-M1, DC/KLH
  Arms: DC/LNCaP

SUMMARY:
The purpose of this study is to assess the safety and activity of a type of vaccine as immune therapy for prostate cancer. This vaccine will be made for each participant's own immune cells (called dendritic cells) obtained by blood donation. Dendritic cells are immune cells, whose role is to identify foreign antigens (bacteria, viruses, or tumor cells, for example) in the body and to activate other cells of the immune system to mount an attack on that foreign antigen. Each participant will be randomized into either Arm 1 (experimental treatment only) or Arm 2 (placebo first, then the experimental treatment). Participants will be given the vaccine and three boosters as an injection. After the placebo phase, each participant in Arm 2 will crossover to the treatment phase so that all participants will eventually receive the experimental treatment.

DETAILED DESCRIPTION:
This is a Phase I/II dendritic cell vaccine study for patients with prostate cancer. Our laboratory has demonstrated that effective tumor immunity in humans is associated with, and likely mediated at least in part by tumor antigen-specific killer T cells (Albert et al., 1998a; Darnell, 1999; Darnell and Posner, 2003). Moreover, we have demonstrated that apoptotic material derived from dying tumor cells are a potent means of delivering antigen to DCs and subsequently triggering tumor antigen-specific T cell responses ex vivo (Albert et al., 1998a; Albert et al., 1998c). In this study, patients with 3 consecutive rises in PSA measured at least 2 week apart, after definite local therapy (prostatectomy or radiation) will be recruited. Peripheral blood monocytes will be collected by leukapheresis and dendritic cells will be generated in the Cleanroom in the Laboratory of Molecular Neuro-Oncology. These dendritic cells will be pulsed with apoptotic prostate cancer cells from a cell line (LNCaP), harvested, tested for certain release criteria, and then injected as vaccine. When patients are found to be eligible for the study, they will be randomized into either the experimental group or the placebo group for the purposes of comparing adverse events between groups only. Vaccine plus 3 boosters (or placebo) will be given, each two weeks apart. After the third booster, patients will be unblinded. Those receiving the vaccine will when enter the follow up phase which includes a post treatment leukapheresis. Those in the placebo group will cross over and receive the vaccine and boosters. The primary outcomes to be evaluated are toxicity and activity. Patients will be evaluated for both local and systemic toxicity. For activity, we measure both immunological and clinical responses to the vaccine, comparing measures taken before and after vaccination, combining patients in both arms.

ELIGIBILITY:
Inclusion Criteria:

Disease Characteristics

* Histologically confirmed prostate carcinoma
* Progressive, disease required, i.e.: elevated PSA documented to be rising on 3 occasions, either despite castrate testosterone levels (below 50 ng/dl), or after definitive local therapy (prostatectomy or radiation).

Prior/Concurrent Therapy

-Biologic therapy:

* Recovered from toxicity of any prior therapy

  -Chemotherapy:
* At least 4 weeks since chemotherapy -Endocrine evaluation/therapy
* 3 rising PSA values at least 2 weeks apart
* At least 2 weeks since concurrent corticosteroids (other than for replacement therapy for adrenal insufficiency)
* Medical hormonal therapy to maintain castrate testosterone levels permitted

  -Radiotherapy:
* At least 4 weeks since radiotherapy

  -Surgery:
* Prior surgery allowed

Patient Characteristics

* Age: 18 and over, able to give written informed consent. Individuals unable to provide informed consent must have consent provided by the legal guardian, or person designated by the subject to give consent on his behalf.
* Performance status: Karnofsky 70-100%
* Life expectancy: At least 1 year
* Hematopoietic: obtained twice, once within 45 days prior to study entry, and again within 72 hours of study entry.
* WBC greater than 3,800
* Absolute neutrophils greater than 1,500
* Absolute lymphocytes greater than 500
* Platelets greater than 120,000
* Hb at least 10 g/dl
* Hepatic:

  --Bilirubin less than 2.0 mg/dl OR

  --SGOT less than 2 x ULN
* Renal:

  * Creatinine no greater than 2.0 mg/dl OR
  * Creatinine clearance at least 40 ml/min
* Rheumatologic:

  --ANA no greater than upper limit of normal, or ANA abnormal in absence of clinical signs of autoimmunity.
  * Rheumatoid factor (RF) no greater than upper limit of normal, or RF abnormal in absence of clinical signs of autoimmunity.
  * Anti-ds DNA no greater than upper limit of normal, or anti ds DNA abnormal in absence of clinical signs of autoimmunity.
* Immunologic:
* Influenza serology (assessment made at time of screening).
* Assessment of DTH response to a standard anergy panel (to include candida, trichophyton and tetanus) or to a Multitest CMI (a disposable kit for DTH testing with standardized preloaded antigens).
* Endocrine:

  --TSH, T3, and T4 no greater than upper limit of normal
* Radiographic:

  * Baseline bone scan
  * Baseline CT or MRI of abdomen and pelvis

Exclusion Criteria:

Disease Characteristics -No active CNS metastases

Prior/Concurrent Therapy

* Biologic therapy:

  * No prior autologous or allogeneic tumor vaccines
  * No concurrent other immunotherapy
* Chemotherapy

  --Not previously treated with more than 2 chemotherapy regimens
  * No concurrent chemotherapy
* Radiotherapy --No concurrent radiotherapy

Patient Characteristics -Cardiovascular: No NYHA class III/IV status No active angina, clinically significant cardiac arrythmia, recent (6 months) myocardial infarction

* Pulmonary:

  --No severe debilitating pulmonary disease
* Other:

  * No active infection requiring antibiotics
  * No active pain requiring chronic opioid analgesics.
  * Not HIV, hepatitis B or hepatitis C virus positive; anti-HIV, HbsAg and Hep C antibody negative
  * No history of hypersensitivity to vaccine components
  * No serious uncontrolled medical illness
  * No currently active second malignancy other than non-melanoma skin cancer (note: a patient is NOT considered to have currently active malignancy if they have completed therapy and are now considered by their physician to be at less than 30% risk for relapse)
  * No history of total lymph node irradiation
  * No history of vasculitis, including but not limited to systemic necrotizing vasculitides (polyarteritis nodosa group), hypersensitivity vasculitis, Wegener's granulomatosis.
  * No history of autoimmune disease.
  * No use of hydroxyurea within 45 days of study entry
  * No receipt of immune modulators or suppressors within 30 days prior to study entry, including but not limited to interferons and thalidomide. No active requirement for corticosteroids; prior use is acceptable.
  * No psychiatric illness or social condition that, in the opinion of the investigator, would interfere with adherence to study requirements.
  * No alcohol or drug use or dependence that, in the opinion of the investigator, would interfere with adherence to study requirements.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2002-03; Primary Completion 2008-11 (Actual); Study Completion 2008-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Robert B. Darnell, MD, PHD, Principal Investigator — Rockefeller University
Locations (1):
- Rockefeller University Hospital, New York, New York, United States

REFERENCES:
- [Derived] Frank MO, Kaufman J, Parveen S, Blachere NE, Orange DE, Darnell RB. Dendritic cell vaccines containing lymphocytes produce improved immunogenicity in patients with cancer. J Transl Med. 2014 Dec 5;12:338. doi: 10.1186/s12967-014-0338-3. PMID 25475068
- [Derived] Frank MO, Kaufman J, Tian S, Suarez-Farinas M, Parveen S, Blachere NE, Morris MJ, Slovin S, Scher HI, Albert ML, Darnell RB. Harnessing naturally occurring tumor immunity: a clinical vaccine trial in prostate cancer. PLoS One. 2010 Sep 1;5(9):e12367. doi: 10.1371/journal.pone.0012367. PMID 20824184

RESULTS

PARTICIPANT FLOW:
Groups:
- Dendritic Cells Pulsed With LNCaP (DC/LNCaP): 12 patients, receiving DC/LNCaP vaccine and the DC/LNCaP-M1 and DC/KLH immunizations over 8 weeks. THE PURPOSE OF THESE 2 ARMS IS TO COMPARE ADVERSE EVENTS (AEs) DURING THE 1ST 8 WKS ONLY.
Period: Overall Study
Arm/Group | Dendritic Cells Pulsed With LNCaP (DC/LNCaP) | Placebo
Started | 12 | 12
Completed | 12 | 12
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Dendritic Cells Pulsed With LNCaP (DC/LNCaP) | Placebo | Total
Number analyzed (Participants) | 12 | 12 | 24
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 5 | 6 | 11
Age Continuous [Mean (Standard Deviation); unit: years] | 62.5 (6.7) | 65.7 (9.2) | 64.0 (7.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 12 | 12 | 24
Region of Enrollment [Number; unit: participants]
  United States | 12 | 12 | 24

OUTCOME MEASURES:

1. Primary Outcome: Adverse Event
Description: Occurrence of adverse events (AE) was compared between the placebo and vaccine groups during the blinded phase (the 1st 9 weeks). At the end of this phase, all were unblinded, and those who received placebo crossed over to now receive vaccine. All serious AEs and any other AEs that occurred 5 times or more are reported. The exact binomial test was used to compare the occurrence of each AE between groups.
Time Frame: End of blinded phase (wk 9)
Population: All AEs occurring 5 or more times during the study were analyzed. All AEs reported are grade 1 except as noted.
Measure: Number; unit: Adverse Events
Groups:
- Placebo: 12 patients receiving vehicle only
Arm/Group | Dendritic Cells Pulsed With LNCaP (DC/LNCaP) | Placebo
Number analyzed (Participants) | 12 | 12
Adverse Events
  injection site reaction | 22 | 2
  injection site reaction (grade 2) | 4 | 0
  albumin, serum, low | 0 | 1
  albumin, urine, high | 2 | 3
  ALT, serum, high | 3 | 4
  ANA, high | 1 | 1
  BUN, serum, high | 4 | 1
  chloride, serum, high | 1 | 4
  CO2 serum, low | 3 | 4
  creatinine, serum, high | 3 | 1
  diarrhea/loose stools | 5 | 1
  edema, lower extremities | 0 | 2
  eosinophils, high | 1 | 3
  fatigue | 6 | 5
  glucose, serum, high, non-fasting | 6 | 5
  ketones, urine, high | 1 | 2
  potassium, serum, high | 0 | 3
  potassium, serum, high (grade 2) | 0 | 1
  rash | 2 | 2
  URI | 3 | 3
  Hospitalization: cardioversion/atrial fibrillation | 1 | 0
Statistical Analysis 1: Comparison: Dendritic Cells Pulsed With LNCaP (DC/LNCaP) vs Placebo; for injection site reaction only; Test type: Superiority or Other; p = 0.001, Fisher Exact
Statistical Analysis 2: Comparison: Dendritic Cells Pulsed With LNCaP (DC/LNCaP) vs Placebo; for all other adverse events; Test type: Superiority or Other; p > 0.2, Fisher Exact

2. Primary Outcome: Immunogenicity of the DC/LNCaP Vaccine. Pre- vs Post-vaccination Bulk T Cell Proliferation (3H Thymidine Incorporation) by Type of Antigen. The "Number" Indicated is the Median Difference of Post-Pre, of Each Antigen Group.
Description: The difference between post minus pre-vaccination bulk T cell proliferation was calculated for each antigen.
Time Frame: pre- vs post-vaccination. Pre-vaccination T cells were collected at Wk 0 and post-vaccination T cells were collected at Wk 13
Population: The Arm/Group Title is different for this outcome. In the 1st outcome analysis, AEs were being compared between placebo and tx groups. After the blinded phase, placebo pts crossover and we compare pre-vs post vaccination T cell proliferation in all pts. 22 of 24 pts'assays were analyzed. Two were excluded as they failed internal controls.
Measure: Median (95% Confidence Interval); unit: cells *10^3 per minute
Groups:
- Median Difference, Post-Pre Vaccination: For each antigen group, the difference between the post and pre-vaccination T cell proliferation response was calculated.
Arm/Group | Median Difference, Post-Pre Vaccination
Number analyzed (Participants) | 22
cells *10^3 per minute
  No Antigen | 4375.64 [-1105.5989 to 10661.4237]
  KLH | 16873.92 [5105.6543 to 28642.1867]
  LNCaP | 20334.1581 [4265.9125 to 36402.4037]
  PC3 | 23950.125 [7006.2329 to 40894.0171]
  Control Antigen (3T3) | 10299.3967 [-777.3295 to 21376.1229]

3. Secondary Outcome: Change in PSA Slope, Pre- vs Post-vaccination.
Description: To model the evolution of PSA (in log-scale) during the three study phases (pre-vaccine, vaccine, and post-vaccine phases), a mixed linear spline model was used. Two knots (one at the start of the vaccine phase and the other at the start of the post-vaccine phase) were used to directly quantify the differences in slopes between each phase. To account for the heterogeneous treatment effect and the repeated measures structure, random effects are incorporated into the model. For the general model, random effects for the intercept, slope and the first knot were considered.
Time Frame: pre- vs post- vaccination PSA slopes.
Population: 23 of 24 patients were analyzed. 1 patient was not evaluable.
Measure: Number (95% Confidence Interval); unit: log₂(ng/ml)/month
Arm/Group | Pre-vs Post-vaccination PSA Slope
Number analyzed (Participants) | 23
log₂(ng/ml)/month | -0.093 [-0.1694 to -0.0166]
Statistical Analysis 1: Comparison: Pre-vs Post-vaccination PSA Slope; Test type: Superiority or Other; p = 0.016, Linear Spline model

ADVERSE EVENTS:
Time Frame: AEs were collected for 29 weeks.
Description: All AEs other than SAEs are Grade 1 (NCI, CTCAE). As this reporting table does not allow having 2 arms initially then 1, all AEs are entered as 1 arm. Specifics for each arm separately is reported in Outcome 1.
Groups:
- Arm 2 Placebo Phase: Single-blind
- Arm 1 Vaccine Phase: Single blind
- Arm 2 Vaccine Phase; Arm 1 and 2 Post-Vaccination Phase: Unblinded
Arm/Group | Arm 2 Placebo Phase | Arm 1 Vaccine Phase | Arm 2 Vaccine Phase | Arm 1 and 2 Post-Vaccination Phase
Serious Adverse Events (participants affected / at risk) | 0/12 | 1/12 | 0/12 | 1/24
Other Adverse Events (participants affected / at risk) | 12/12 | 12/12 | 12/12 | 22/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs (number of events):
Term (organ system) | Arm 2 Placebo Phase (N=12) | Arm 1 Vaccine Phase (N=12) | Arm 2 Vaccine Phase (N=12) | Arm 1 and 2 Post-Vaccination Phase (N=24)
Elective Hospitalization: inguinal hernia repair (Surgical and medical procedures) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
Elective Hosptalization: cholecystectomy (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Hospitalization: cardioversion for atrial fibrillation (Cardiac disorders) | 0/0 (0) | 1 (1) | 0 (0) | 0 (0)
Hospitalization: urinary retention (Renal and urinary disorders) | 0/0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm 2 Placebo Phase (N=12) | Arm 1 Vaccine Phase (N=12) | Arm 2 Vaccine Phase (N=12) | Arm 1 and 2 Post-Vaccination Phase (N=24)
ALT, serum, high (General disorders) | 3 | 2 | 1 | 2 (2)
ANA (General disorders) | 1 | 1 | 3 | 4
BUN, serum, high (General disorders) | 1 | 3 | 2 | 1
CO2, serum, low (General disorders) | 4 | 2 | 2 | 1
URI (Respiratory, thoracic and mediastinal disorders) | 3 | 3 | 1 | 0
albumin, serum, low (General disorders) | 0 | 1 | 3 | 0
albumin, urine, high (General disorders) | 1 | 3 | 0 | 3
chloride, serum, high (General disorders) | 4 | 1 | 0 | 2
creatinine, serum, high (General disorders) | 1 | 2 | 2 | 2
diarrhea/loose stools (Gastrointestinal disorders) | 1 | 3 | 0 | 0
edema, lower extremities (General disorders) | 2 | 0 | 1 | 1
eosinophils, high (Blood and lymphatic system disorders) | 3 | 1 | 1 | 1
fatigue (General disorders) | 5 | 5 | 4 | 0
glucose, serum, high, non-fasting (General disorders) | 5 | 6 | 1 | 6
ketones, urine, high (Renal and urinary disorders) | 2 | 1 | 1 | 3
potassium, serum, high (General disorders) | 4 | 0 | 5 | 1
rash (Skin and subcutaneous tissue disorders) | 2 | 1 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No